CLINICAL TRIAL: NCT05643833
Title: Impact of Gender on the Outcome of Liver Transplantation for Hepatocellular Carcinoma: A Multicenter Retrospective Study in China
Brief Title: Impact of Gender on the Outcome of Liver Transplantation for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2022-ZJU-OBS1
Record Dates: First submitted 2022-11-29; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Cancer of Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Male recipient
  Interventions: Other: no intervention
- Female recipient
  Interventions: Other: no intervention
- Male donor
  Interventions: Other: no intervention
- Female donor
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This is a large-scale study in China to provide evidence and insights in the role of gender in LT for HCC by analyzing the data of 3769 recipients with HCC registered in the China Liver Transplant Registry.

ELIGIBILITY:
Inclusion Criteria:

The patients with liver transplants performed from January 2015 to December 2020, whose clinicopathological data were registered in the CLTR.

Exclusion Criteria:

Patients with following features were excluded: with concurrent other malignancies, pathologically-confirmed tumor types other than HCC, such as intrahepatic cholangiocarcinoma (ICC), combined hepatocellular cholangiocarcinoma (cHCC-CC), fibrolamellar hepatocellular carcinoma (FLC) or secondary metastatic tumor; without histological confirmation of HCC for transplantation. The patients who received living donor liver transplantation, split liver transplantation, reduced-size liver transplantation or simultaneous transplantation were also excluded. Next, pediatric patients (<18 years) or senile patients (>65 years) and those patients who died within six months after transplantation were also excluded. Finally, the patients with type-1 and type-2 portal vein tumor thrombus (PVTT), tumor metastasis, having doubtful or contradictory data or missing essential data for analysis, re-transplantation during follow-up time were excluded as well.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 3769 HCC patients underwent liver transplant with the age between 18-65 years old were studied.
Sampling Method: Probability Sample
Enrollment: 3769 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | January 2015 to December 2020
  the overall survival of liver transplant recipient with HCC

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No